CLINICAL TRIAL: NCT02025868
Title: Systematic "Adherence Intervention" Phase Before Switching to 3rd-line ART in Patients With 2nd-line ART Virologic Failure in Sub-Saharan Africa : a Phase 2b Non-randomized Study.
Brief Title: Third Line Antiretroviral Treatment Optimization in Sub-Saharan Africa
Acronym: THILAO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12269 THILAO
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: HIV Infection
Keywords: Africa; Antiretroviral Treatment; Adherence reinforcement; Third line ART; Second line ART; Virologic failure; Adults
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adherence reinforcement before switch to 3rd-line ART (Experimental)
  Interventions: Behavioral: adherence reinforcement; Drug: Antiretroviral Therapy Darunavir/r + Raltegravir + 2 NRTIs (as chosen by the investigators)

INTERVENTIONS:
Behavioral: adherence reinforcement — Directly observed treatment at home (family or relatives DOT); pillboxes; phone calls; SMS; home visits; adherence reinforcement sessions by trained health workers.
Drug: Antiretroviral Therapy Darunavir/r + Raltegravir + 2 NRTIs (as chosen by the investigators) — Second-line ART regimen : ongoing regimen at the time of inclusion will be continued.
  Third-line ART regimen : Darunavir/r + Raltegravir + 2 NRTIs (as chosen by the investigators)

SUMMARY:
Thilao is a multi-country, phase 2b, non-randomized study, in Burkina Faso, Cote d'Ivoire, Mali and Senegal, West Africa.

HIV-1 adults with 2nd-line ART virologic failure (plasma HIV-1 RNA >1000 copies/ml) will be recruited and followed in two phases:

* First, a 12-week intentive adherence reinforcement phase, during which patients will continue 2nd-line ART, be seen repeatidly for counseling and educational training on adherence, and be offered the possibility of phone, SMS and home visit contacts with social workers;
* Second, a 48-week phase, during which:

  * Patients successfully resuppressed at the end of the first phase will continue 2nd-line ART and adherence reinforcement;
  * Patients with persitent virologic failure will switch to a darunavir/r + raltegravir-based 3rd-line ART.

Genotype resistance tests will be performed retrospectively on frozen samples. The main outcome will be the percentage of patients with plasma HIV-1 viral RNA <50 copies/ml at 64 weeks.

DETAILED DESCRIPTION:
Main objective

To estimate, in sub-Saharan African HIV-1 infected adults who failed a NNRTI-base first-line ART and then a PI-based second-line ART:

1. The efficacy (and associated factors) at 12 weeks of an intensive 3-months adherence reinfrocement phase;
2. In patients who successfully resuppress at 12 weeks: The percentage of patients still with continuing succesfull virologic supression on 2nd-line ART at 64 weeks (and factors associated to success) ;
3. In patients with persistent failure at 12 weeks : The efficacy (and associated factors) at 64 weeks of a darunavir/r + raltegravir-based 3rd-line regimen.

Number of participants : 200

Main outcome :

* At 12 weeks : Proportion of patients with a plasma HIV-1 RNA <400 copies/ml and/or with a decrease in plasma HIV-1 RNA >2 log10 copies/ml between inclusion and 12 weeks;
* At 64 weeks : proportion of patients with a plasma HIV-1 RNA <50 copies/ml.

Inclusion criteria:

* Age >18 years
* Documented HIV-1 infection.
* History of failing a NNRTI-based 1st-line ART
* Current PI-based 2nd-line ART >6 months
* Plasma HIV-1 RNA >1000 copies/ml
* Signed informed consent

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Documented HIV-1 infection
* History of failing a NNRTI-based 1st-line ART
* Current PI-based 2nd-line ART >6 months
* Plasma HIV-1 RNA >1000 copies/ml
* Signed informed consent

Exclusion Criteria:

* HIV-2 infection
* Any Severe clinical event under exploration
* History of treatment including darunavir or raltegravir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Virologic efficacy of the adherence reinforcement intervention | Week 12
  Proportion of patients with plasma viral load <400 copies/ml at Week 12 and/or with a decrease in plasma viral load >2 log10 copies/ml between inclusion and Week 12
Persistent virologic efficacy of the adherence reinforcement intervention | Week 64
  Proportion of patients with plasma viral load <50 copies/ ml at Week 64 among those who stayed on 2nd-line ART at Week 16
Virologic efficacy of 3rd-line ART | Week 64
  Proportion of patients with HIV-1 plasma viral load <50 copies/ml at Week 64 among those with persistent failure at Week 12 who switched to 3rd-line ART

SECONDARY OUTCOMES:
Immunological efficacy of the adherence reinforcement intervention | Week 12
  CD4 count evolution between inclusion and Week 12
Immunological efficacy of 3rd-line ART | Week 64
  CD4 count evolution between Week12 and Week 64 among patients who switched to 3rd-line ART at Week 16
Tolerance of 3rd-line ART drugs | Week 64
  Incidence of grade 3-4 adverse events (ANRS grading table) in patients on 3rd-line ART
Adherence to 3rd-line ART | Week 64
  3rd-line Medication Possession Ratio between Week 16 and Week 64
Resistance to 1st and 2nd-line antiretroviral drugs | Week 12
  Resistance mutations to antiretroviral drugs among patients with virological failure at Week 12
Resistance to 1st, 2nd and 3rd-line antiretroviral drugs | Week 64
  Resistance mutations to antiretroviral drugs among patients with virological failure at Week 64
Plasma antiretroviral drugs concentration | Week 12
  Plasma antiretroviral drugs concentration at Week 12
Plasma antiretroviral drugs concentration | Week 64
  Plasma antiretroviral drugs concentration at Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Serge P. Eholie, MD, MSc, Pr, Principal Investigator — Service des Maladies Infectieuses et Tropicales, CHU de Treichville, Abidjan, Côte d'Ivoire; Roland Landman, MD, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Hôpital Bichat Claude Bernard, Paris, France; Xavier Anglaret, MD, PhD, Study Director — Inserm 897, University of Bordeaux, France; Pierre-Marie Girard, MD, PhD, Study Chair — Infectious Diseases Department, University Hospital Saint Antoine, Paris, France
Locations (7):
- Burkina Faso (2):
  - CHU Sourô Sanou, Bobo-Dioulasso
  - CHU Yalgado Ouedraogo, Ouagadougou
- Côte d’Ivoire (2):
  - Centre de Prise en Charge et de Formation (CePReF), Association ACONDA, Abidjan
  - Service des Maladies Infectieuses et Tropicales (SMIT), Abidjan
- Mali (2):
  - Centre d'Ecoute, de Soins, d'Animation et de Conseils (CESAC), Bamako
  - CHU Point G, Bamako
- CHU Fann, Dakar, Senegal

REFERENCES:
- See also: Sponsor site — http://anrs.fr/
- See also: Related Info — http://www.mereva.net/